CLINICAL TRIAL: NCT06574308
Title: Clinical Evaluation of the Scopio Cell Morphology Technology on Pre-classification of Blood Cells in Peripheral Blood (PB) and Bone Marrow (BM)
Brief Title: Clinical Evaluation of the Scopio Cell Morphology Technology
Acronym: Hemascopio
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6901
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Blood Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood cells classification — Comparison of the classification of peripheral blood and bone marrow cells with optical microscope reading with pre-classification using Scopio technology (AI based)

SUMMARY:
Digital morphology is currently expanding and developing new applications based on artificial intelligence software. We recently published a study comparing screen validation and microscopic reading of bone marrow aspirates. The aim of the current research will be the comparison between optical microscope reading and automatic pre-classification (AI based)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from hemopathies with bone marrow aspirate assessable under the optical microscope

Exclusion Criteria:

* Patients not affected by blood disorders
* Patients suffering from hemopathies with bone marrow aspirate that cannot be assessed under the optical microscope

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pazienti affetti da emopatie
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Optical microscope reading and automatic pre-classification | 12 months
  Comparison between optical microscope reading and automatic pre-classification (AI based)

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Chiusolo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy